CLINICAL TRIAL: NCT03115554
Title: Comparison of Pulmonary Vein Isolation Plus Additional Catheter Ablation or Pulmonary Vein Isolation Alone for the Treatment of Atrial Fibrillation for Patients With Paroxysmal Atrial Fibrillation: A Prospective, Randomized Study
Brief Title: Comparison of PVI Plus Catheter Ablation or PVI Alone for the Treatment of AFib for Patients With Paroxysmal Atrial Fibrillation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients did not want to be randomized in their procedure.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-74
Record Dates: First submitted 2017-03-13; First posted 2017-04-14 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2017-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI Plus Catheter Ablation (Active Comparator): Patients with sustained AF following PVI will receive additional linear or focal intracardiac catheter ablation for AF.
  Interventions: Procedure: PVI Plus Catheter Ablation
- PVI Alone (Active Comparator): Patients with sustained AF following PVI will not receive additional linear or focal intracardiac catheter ablation for AF.
  Interventions: Procedure: PVI Alone

INTERVENTIONS:
Procedure: PVI Plus Catheter Ablation — Patients with sustained AF following PVI will receive additional linear or focal intracardiac catheter ablation for AF.
  Arms: PVI Plus Catheter Ablation
Procedure: PVI Alone — Patients with sustained AF following PVI will not receive additional linear or focal intracardiac catheter ablation for AF.
  Arms: PVI Alone

SUMMARY:
There is a need to compare the efficacy of PVI versus PVI plus catheter ablation, which includes ablation of complex fractionated atrial electrograms (CFAE) and linear lesions in the same procedure. If it is found that the PVI alone is as effective as PVI plus catheter ablation of CFAE and linear lesions, it may reduce the need for catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

(Step 1 - Registration)

* The subject is 18 years of age or older
* Left atrium < 6.0 cm (Trans Thoracic Echo - TTE - parasternal 4 chamber view
* performed within 6 months)
* Documentation of AF that terminates spontaneously or with intervention within 7 days of onset (PAF) Failed or refractory to one AAD (class I and/or III)
* Provided written informed consent
* Be eligible for an AF ablation procedure for Paroxysmal AF

(Step 2 - Randomization)

* Sustained AF following PVI with ability to receive additional linear or focal intracardiac catheter ablation

Exclusion Criteria:

(Step 1 - Registration)

* Pregnant or planning to become pregnant during study
* Co-morbid medical conditions that limit one-year life expectancy
* Previous cardiac surgery
* Patients who have active infection or sepsis
* Patients with esophageal ulcers strictures and varices
* Patients who are contraindicated for anticoagulants such as heparin and warfarin
* Patients who are being treated for ventricular arrhythmias
* Patients who have had a previous left atrial catheter ablation for AF (does not
* include ablation for AFL or other supraventricular arrhythmias)
* Current participation in another clinical investigation of a medical device or a drug, or recent participation in such a study within 30 days prior to study enrollment
* Not competent to legally represent him or herself (e.g., requires a guardian or
* caretaker as a legal representative)

(Step 2 Randomization)

* Not able to receive additional linear or focal intracardiac catheter ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
Time to recurrence | 12 months
  Any atrial fibrillation/atrial tachycardia/atrial flutter following the blanking period.

SECONDARY OUTCOMES:
Time to recurrence following intervention | 12 months post intervention
  Time to recurrence following intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jasbir Sra, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora Health Care, Milwaukee, Wisconsin, United States